CLINICAL TRIAL: NCT04165356
Title: Efficacy of Mouth-rinse With Chlorhexidine for the Prevention of Ventilator-associated Infections in Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autónoma de Yucatán (Other)
Collaborators: Hospital Regional de Alta Especialidad de la Península de Yucatán (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-013
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infections Associated With Mechanical Ventilation; Pneumonia Associated With Mechanical Ventilation
Keywords: Chlorhexidine mouthwashes; chlorhexidine efficacy; artificial respiration; cross infection; ventilator-associated pneumonia
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated | interventions — Mouthwashes; Isotonic Solutions; Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: Randomly asignated to one of two parallel groups of mouth-rinse treatments:
  1. Mouth-rinse with 0.12% clorhexidine + tooth brushing twice daily
  2. Mouth-rinse with isotonic solution with 1.5% sodium bicarbonate + tooth brushing twice daily
Who Masked: Participant, Care Provider
Masking Description: All mouth-rinse bottles will have the same external appearance, being plastic bottles with integrated spray atomizer and protective plastic cap. Each bottle will have a unique folio for identification printed on the identification label.
  The clinical staff working in the Hospital and having contact with the study subjects will be blinded at all times to the care group assigned to the patient.
  Academic staff working outside the Hospital and will not have direct contact with the study subjects, will not be blinded to the assigned group, in order to administer a second bottle of treatment if necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mouth-rinse with clorhexidine (Experimental): Mouth-rinse with 0.12% clorhexidine + tooth brushing twice daily
  Interventions: Procedure: Mouth-rinse with 0.12% clorhexidine
- Mouth-rinse with bicarbonate isotonic solution (Active Comparator): Mouth-rinse with isotonic solution with 1.5% sodium bicarbonate + tooth brushing twice daily
  Interventions: Procedure: Mouth-rinse with isotonic solution with 1.5% sodium bicarbonate

INTERVENTIONS:
Procedure: Mouth-rinse with 0.12% clorhexidine — mouthwash with 0.12% chlorhexidine twice daily compared to isotonic bicarbonated solution twice daily for the prevention of any infection associated with mechanical ventilation in patients requiring endotracheal intubation in the intensive care unit of a third level hospital.
  Arms: Mouth-rinse with clorhexidine
Procedure: Mouth-rinse with isotonic solution with 1.5% sodium bicarbonate — mouthwash with sotonic solution with 1.5% sodium bicarbonate twice daily for the prevention of any intection associated with mechanical ventilation
  Arms: Mouth-rinse with bicarbonate isotonic solution

SUMMARY:
Background:

Infections associated with mechanical ventilation are associated with high rates of morbidity and mortality, which results not only in an increase in hospitalization days and care costs, but also in an increase in DALYS (years of life disability adjustment) in the population.

Critically ill patients have a high risk of infection as a result of underlying immunodeficiency, comorbidity and placement of invasive devices (such as endotracheal tubes and intravascular devices). Infections in these patients constitute a challenge for hospital authorities, as they are considered a social and economic problem that influences the quality of care, in a system where health services are increasingly affected by high patient care costs and the reduction of public spending.

The decrease in the number of bacteria in the oral cavity reduces the presence of microorganisms available for translocation and colonization of the lower respiratory tract; Therefore, performing oral care intervention is considered an economically attractive method to reduce the risk of developing infections associated with endotracheal intubation.

In our environment, oral cleaning is performed as part of the nursing care package granted to all patients of the ICU, however, there is no standardized method among nursing staff that guarantees the desired prevention.

Objective: To evaluate the efficacy and safety of mouth-rinse with 0.12% chlorhexidine to prevent infections associated with mechanical ventilation in patients in the intensive care unit in a third level hospital in Mérida, Yucatán.

Hypothesis: Mouth-rinse with 0.12% chlorhexidine twice daily more effective and safe than mouthwash with bicarbonated isotonic solution twice daily to prevent infections associated with mechanical ventilation in patients in the intensive care unit of a hospital third level.

Methodology: Double-blind randomized controlled clinical trial with active substance for the evaluation of the non-inferiority of the efficacy and safety of mouthwash with 0.12% chlorhexidine twice daily compared to isotonic bicarbonated solution twice daily for the prevention of any infection associated with mechanical ventilation in patients requiring endotracheal intubation in the intensive care unit of a third level hospital.

DETAILED DESCRIPTION:
Eligibility criteria Adult patients admitted to the ICU will be included, with less than 24 hours of endotracheal intubation due to mechanical ventilation requirements, whose responsible family member gives informed consent.

Patients with known hypersensitivity or contraindications for the use of oral chlorhexidine, patients with a diagnosis of admission to the ICU of any respiratory tract infection, toothless patients and pregnant patients will be excluded.

Patients who, during their stay in ICU, require tracheostomy after having endotracheal intubation and those who decide to withdraw their informed consent will be eliminated from the active phase.

Adverse events surveillance During the period of the permanence of the subject in the clinical trial, daily monitoring of adverse events and the response variable will be carried out, taking information from the clinical record, the results of cultures performed on the patient and supplemented with hospital surveillance reports.

Treatment assignation According to the randomization of the subject, a bottle of mouthwash labeled with the clinical trial data will be assigned for personal use.

The said bottle may correspond to one of two treatments:

1. Mouth-rinse with 0.12% chlorhexidine, 35 ml spray bottle, with a capacity of 200 shots, Clorhex-gum® brand.
2. Mouth-rinse with an isotonic solution with 1.5% sodium bicarbonate, 35ml spray bottle, with a capacity of approximately 200 shots.

All mouth-rinse bottles will have the same external appearance, being plastic bottles with integrated spray atomizer and protective plastic cap. Each bottle will have a unique folio for identification printed on the identification label.

The mouthwash bottles will be stored in the hospital area, under the shelter of the participating clinical staff, in a cool, dark and locked space.

Once the vial has been assigned to a patient, it will remain next to the subject's bed for the sole and individual use of the said subject.

Blind and no blind staff The investigators, that will be in contact with patients, will be blinded at all times to the care group assigned to the patient.

Intention to treat analysis The analysis of the subjects participating in the clinical trial will be performed according to the treatment group to which they were randomized, regardless of whether they completed the study procedures, adherence to established care or follow-up time.

Dependent variable The response variable will be the incidence rate of infections associated with Mechanical Ventilation (whose denominator will be the observation time in person-days) developed during the period of the permanence of endotracheal intubation and up to 48 hours after withdrawal (or death). of the patient).

The IAVM that will be searched intentionally are:

* Pneumonia Associated with Mechanical Ventilation
* Bronchitis or bronchitis trachea
* Laryngitis
* Bacterial pharyngitis
* Acute sinusitis

Mouth-rinse procedure During the active phase: Every 12 hours, approximately, the oral antiseptic decontamination of the study subjects will be carried out, at the time in which secretions will be aspirated.

According to the recommendations of the Clorhex-gum® data sheet (see annex 1) and the recommendations for oral hygiene in intubated patients, the procedure to be implemented will be as follows:

1. Hand washing and non-sterile gloves footwear.
2. Exam of the pneumotrop pressure, minimizing the possibility of micro aspirations during the procedure.
3. Removal the may or bite tube, if applicable.
4. Hand washing and sterile globes footwear
5. Aspiration endotracheal and oropharyngeal secretions.
6. Application of approximately 15 shots to cover teeth, mucous membranes and tongue.
7. Tooth brushing (Using the brush that will be delivered at randomization) to remove the interdental bacterial plaque.
8. After 2 to 3 minutes, aspiration of the remnants of the rinse with a sterile atraumatic probe to gently aspirate
9. Removal the endotracheal tube holder.
10. Dried up lips and the surrounding area, while checking out the condition of the corners of the mouth and mucous membranes.
11. Change the position of the endotracheal tube (holding it with a clean fixation)
12. Application of lip protection
13. Placement the may tube or bite, if necessary.

Dental plaque cultures

As part of the study procedures, 2 dental plaque cultures are contemplated during the course of the study, which will be carried out by trained clinical staff, following the following recommendations:

* They must be performed under conditions of maximum asepsis, avoiding environmental contamination, medical personnel and the patient himself.
* The sample should not be in contact with disinfectant substances, so it must be done before oral hygiene.
* The request handout and sample identification must follow the characteristics requested by the hospital laboratory.
* The sample will be taken with the use of curettes and swabs of the dental plaque, trying to cover in the margin of the gum, both in the upper and lower jaw.
* The sample will be stored at room temperature and analyzed with the standard procedure.

Statistic analysis A descriptive statistical analysis will be carried out to detail the sociodemographic and clinical characteristics of the subjects belonging to both oral care groups. The proportions of the variables of both groups will be compared using chi-square tests, while the differences in the means will be evaluated through the Student's T-test.

The cumulative incidence of infections associated with mechanical ventilation and pneumonia associated with mechanical ventilation, between both care groups will be determined and a comparative analysis will be carried out between the different types of infections developed during the period of the permanence of endotracheal intubation and up to 48 hours after withdrawal or until the patient's death. The numerator will be the total of each type of IAVM diagnosed and the denominator will be the sum of individual observation times. The Relative Risk will be calculated from the Incidence Rates and the Population Preventable Fraction for each type of IAVM analyzed.

The Kaplan-Meyer estimator will be used to compare the cumulative curves of days in ICU free of infections associated with mechanical ventilation between care groups with 0.12% chlorhexidine mouthwash and isotonic bicarbonate solution. The potential weights assumed by each oral care group will be compared using the Log Rank test against the incidence rate of infections associated with MV.

As a multivariate analysis, a Poisson regression model will be carried out to determine the effect of 0.12% chlorhexidine mouthwash on the development of IAVM, compared to mouthwash with bicarbonate isotonic solution, in adults hospitalized in intensive care that require mechanical ventilation. adjusting for confusing variables.

To analyze the changes in the dental plaque of the subjects of the two care groups reported in the 3 cultures performed (on day 0, at 24-48hrs and in extubation), a fixed-effects model of analysis of variance For all analyzes a 95% confidence interval and a significance level of p <0.05 will be considered. The analysis will be carried out in the statistical package STATA 14.0 (Stata Corp, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU will be included, with less than 24 hours of endotracheal intubation due to mechanical ventilation requirements, whose responsible family member gives informed consent.

Exclusion Criteria:

* Patients with known hypersensitivity or contraindications for the use of oral chlorhexidine, patients with a diagnosis of admission to the ICU of any respiratory tract infection, toothless patients and pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Infections Associated with Mechanical Ventilation. | Developed during the period of permanence of endotracheal intubation procedure and up to 48 hours after its withdrawal
  New cases of respiratory infections (except pneumonia) developed in susceptible individuals entering the study, during the period of the study.
Cumulative incidence of Pneumonia Associated with Mechanical Ventilation | Developed during the period of permanence of endotracheal intubation procedure and up to 48 hours after withdrawal
  New cases of pneumonia associated with mechanical ventilation developed in susceptible individuals entering the study, during the period of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Rosado Alcocer, MPH, Principal Investigator — Facultad de Enfermería, Universidad Autónoma de Yucatán
Locations (1):
- Hospital Regional de Alta Especialidad de La Peninsula de Yucatan, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No